CLINICAL TRIAL: NCT06420427
Title: Dynamic Monitoring of Circulating Tumor DNA (ctDNA) and HPV DNA in Plasma for the Early Prediction of Recurrence After Cervical Cancer Surgery/Treatment
Brief Title: Dynamic Monitoring of ctDNA and HPV DNA in Plasma for the Early Prediction of Recurrence After Cervical Cancer Surgery
Status: Recruiting | Type: Observational
Sponsor: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Sheng Xiujie, Professor, The Third Affiliated Hospital of Guangzhou Medical University
Other Study IDs: CCA2024005
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: cfHPV DNA in Plasma of Cervical Cancer Patients
Keywords: cfHPV DNA; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Assess the risk of recurrence and the efficacy of medication — Evaluation of recurrence risk and medication efficacy through liquid biopsy

SUMMARY:
Assess the sensitivity, specificity, positive predictive value, and negative predictive value of dynamic monitoring of circulating tumor DNA (ctDNA) combined with circulating HPV DNA (cfHPV DNA) for early prediction of recurrence in cervical cancer post-surgery or post-treatment, and compare its advantages and disadvantages with existing diagnostic methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed HPV-positive cervical malignancy at stages I-IV who have not undergone surgery, radiation therapy, or chemotherapy.
* Patients must be older than 18 years of age.
* Cervical cancer patients who are eligible for surgery and/or chemoradiotherapy.
* Estimated life expectancy of more than three months.
* Understands the study protocol and voluntarily participates in the research by signing the informed consent form.
* Able to provide specimens and corresponding clinical information at each time point.

Exclusion Criteria:

* Patients who are participating in other clinical trials.
* Pregnant or breastfeeding women.
* Patients with severe mental illness.
* Patients who voluntarily withdraw.
* Patients unable to complete the study protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with newly diagnosed HPV-positive cervical malignancy at stages I-IV who have not undergone surgery, radiation therapy, or chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
sensitivity | 2 year
  true positive rate

CONTACTS AND LOCATIONS:
Overall Officials: Xiujie Sheng, Prof, Study Chair — The Third Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
publish an article